CLINICAL TRIAL: NCT06512038
Title: A Pilot Study of the Use of Dual-Energy X-ray Absorptiometry (DXA) in Scoliosis
Brief Title: The Use of DXA in Scoliosis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sheffield Children's NHS Foundation Trust (Other)
Collaborators: University of Sheffield (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 335664
Record Dates: First submitted 2024-05-08; First posted 2024-07-22 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: Scoliosis Idiopathic
Keywords: scoliosis; Juvenile Scoliosis; Adolescent Scoliosis
MeSH Terms: conditions — Scoliosis | interventions — Absorptiometry, Photon

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ADDITIONAL DEXA SCAN (Other): There is only 1 arm on this trial, if a participant agrees to take part they will have additional DEXA radiograph.
  Interventions: Radiation: DEXA Scan

INTERVENTIONS:
Radiation: DEXA Scan — If the participant consents to take part in the trial, they will have an additional DEXA scan.

SUMMARY:
This is a pilot study to look at image quality of iDXA AP supine spinal images to see if the investigators can accurately measure the size of the curve from iDXA images and to see how patients with scoliosis feel about iDXA imaging compared to normal x-rays. With normal x-rays being taken standing (or sitting if patients are in a wheelchair), it is important that the investigators understand how the lying down images compare to the standing images. Where there may be some clinical benefit, images will be taken standing (normal x-rays) and lying down (iDXA images). The investigators will see if the addition of iDXA images can help in brace design and brace monitoring.

DETAILED DESCRIPTION:
This pilot study is an interventional study where patients having routine standing or sitting spinal x-rays for scoliosis monitoring or as part of a treatment protocol will be approached to see if they would have an additional supine AP DXA image. Participants will only have one additional DXA image during the pilot study. The consent will be obtained by one of the spinal surgeons or a specialist spinal nurse. The DXA scan will be performed by one of the radiographers. This study may be performed by a medical student or junior doctor (either would be part of the care team) and supervised by the PI.

The pilot study is expected to last 9 months and consist of 25 patients. The DXA images will be reviewed by 2 consultant spinal surgeons and a consultant radiologist who will make a collective decision every month as to whether the study, or that part of the study, should continue.

Two scoliosis patients have read the study protocol and given their input. The Sheffield Children's Hospital Scoliosis PPI group will feedback on key aspects during the study and help define future studies suggested by this study.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Adolescent Idiopathic Scoliosis (AIS, aged 10-16 years) or Juvenile Idiopathic Scoliosis (JIS, aged 4-9 years) having an x-ray to look for curve progression OR to guide design of a new brace.
* Patients with quadriplegic Cerebral Palsy (CP) having an x-ray to look for curve progression. Within the age range for inclusion for patients with CP, the recruiting clinician will make a clinical judgement on whether the patient is able to lie still long enough to undertake the iDXA, before inviting the patient to take part.

Exclusion Criteria:

* Parents unable to understand the study procedures.
* Patients unable to lie still for 1-2 minutes

Ages: 4 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2024-05-08 (Actual); Primary Completion 2024-12-06 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Radiation Dosage | Through study completion, an average of 6 months
  DXA in comparison to X-Ray
Patient Satisfaction Questionnaire about the use of DXA in Scoliosis | through study completion, an average of 6 months
  This will be self reported questionnaire completed by patients. They will use a simple pictorial scale to report about their experiences having both a DXA and X-ray. The Scale ranges from 'Very Uncomfortable/ very unacceptable', 'Uncomfortable / unacceptable' to 'Okay'.
DXA Image Quality | Through study completion, an average of 6 months
  Image quality as judged by 2 spinal surgeons and a consultant radiologist on a 4 point scale as:
  1. Excellent - almost as good as an x-ray
  2. Good - Good quality and easily able to see required anatomical landmarks for measurement
  3. Adequate - Poor quality but just able to see required anatomical landmarks for measurement
  4. Poor - Unable to see required anatomical landmarks for measurement
Imaging Angles | Through study completion, an average of 6 months
  Cobb angle, apical vertebral translation and apical vertebral rotation will be measured from the x-rays and DXA scans for all the curves
Beighton Score for joint flexibility | Through study completion, an average of 6 months
  Beighton score (flexibility) will be recorded by a clinician for all the patients with idiopathic scoliosis. The score will evaluate each patient's:
  * Passive dorsiflexion and hyperextension of the fifth MCP joint beyond 90°
  * Passive apposition of the thumb to the flexor aspect of the forearm
  * Passive hyperextension of the elbow beyond 10°
  * Passive hyperextension of the knee beyond 10°
  * Active forward flexion of the trunk with the knees fully extended so that the palms of the hands rest flat on the floor

CONTACTS AND LOCATIONS:
Locations (1):
- Sheffield Children's NHS Foundation Trust, Sheffield, United Kingdom

IPD SHARING:
Plan to Share IPD: No